CLINICAL TRIAL: NCT04295304
Title: Safety and Performance Evaluation of the NR600 System in Subjects With End-stage Inherited Outer Retinal Degenerative Diseases
Brief Title: NR600 System Retinal Prosthesis for Patients With Retinal Degenerative Diseases
Acronym: NR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Nano Retina (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NR-DOC-14670
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Retinitis Pigmentosa; Retinal Degeneration
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NR600 device implantation (Experimental): Retinal surgery and implantation of epi-retinal prosthesis
  Interventions: Device: Retinal surgery with implantation of epi-retinal device

INTERVENTIONS:
Device: Retinal surgery with implantation of epi-retinal device — Retinal surgery and implantation of epi-retinal prosthesis

SUMMARY:
The study objective is to demonstrate safety of the NR 600 System, and to evaluate the performance of the device in restoring visual activity of daily living in subjects with retinal degenerative diseases and severe visual impairment

DETAILED DESCRIPTION:
The NR600 is a retinal prosthetic system intended to provide electrical stimulation to the retina to induce visual perception in patients with severe to profound vision loss due to degenerative retinal disease. The system is consisting of an autonomous epiretinal implant with penetrating electrodes, Glasses and a Clinician Station. The implant is Infrared (IR) powered and is designed to convert visual input into well-defined electrical stimulation patterns suited to elicit neuronal retina activity. All study subjects will be implanted with the device in one eye and will be followed for 18-months.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed diagnosis of end-stage hereditary outer retinal degeneration such as RP or cone-rod dystrophy
* Visual acuity in both eyes from light perception to no light perception
* Confirmed functional ganglion cells and optic nerve in the implanted eye
* History of useful vision
* Mentally competent

Exclusion Criteria:

* Diseases or condition that affect retinal and or optic nerve function
* Optic Nerve diseases
* Diseases or conditions that, in the judgement of the surgeon, impede the ability to implant the device or would prevent the system from functioning
* Dry eye
* Pre-disposition to eye rubbing
* Posterior pole severe staphyloma
* Strabismus superior to 10 prismatic diopter
* Severe nystagmus
* Corneal endothelium density < 1500 cells/mm2
* Refractive error ≥±8 diopters spheric and 3.5 diopter cylindric
* Currently pregnant (female subject) or inadequate contraceptive treatment in female subjects <50 years of age.
* Hyperthyroidism or hypersensitivity to iodine
* Neurological and/or psychiatric diseases (e.g. M. Parkinson, epilepsy, depression)
* Participation in another study with any investigational drug or device that may conflict with the objectives, follow-up or testing of this study
* Conditions likely to limit life to less than 1 year from time of recruitment to the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Safety endpoint | within 9 months post implantation
  Occurrence of serious adverse events related to the device and/or to the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Weinberger Dov, Prof., Study Chair — Retinal surgeon
Locations (6):
- Belgium (2):
  - UZ Ghent, Ghent
  - UZ Leuven, Leuven
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
- Italy (2):
  - San Raffaele, Milan
  - Fondazione Policlinico A. Gemelli, IRCCS, Rome

IPD SHARING:
Plan to Share IPD: No